CLINICAL TRIAL: NCT01395511
Title: Acupuncture for Whiplash Associated Disorder: a Randomised, Waiting-list Controlled, Open-label, Parallel-group Pilot Trial
Brief Title: Acupuncture for Whiplash Associated Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: University of Tsukuba (Other)
Responsible Party: Do-Young Choi, Department of Acupuncture & Moxibustion, Kyunghee Oriental Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOMC MIRB2009-05
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2009-12

CONDITIONS: Whiplash Associated Disorder (WAD)
Keywords: whiplash associated disorder,; Intractable Traumatic Cervical Syndrome,; Acupuncture,; Randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): About ten acupuncture points are selected from the following points to be used. Local Acupoints : SI14, SI15, BL10, BL12, BL13, BL14, TE15, GB20, SI9
  Distal Acupoints :
  * Upper extremities: LU6, LU7, LU9, LI11, HT3, SI2, SI3, SI5, SI7, PC4, PC6, TE5
  * Lower extremities: SP3, SP4, BL59, BL60, BL61, BL62, BL66, KI3, KI4,KI6, KI7, GB40, GB41, LR4
  All Acupuncture points were prepared with 70% alcohol pads, and disposable stainless steel needles were used. Most of acupuncture were inserted vertically 1~1.5cm in depth until patient can feel De-Qi. (No more additional stimulation)
  Interventions: Device: Acupuncture
- Waiting list group (No Intervention): No Intervention Comparator
  The waiting-list group did not receive acupuncture treatment and participants were permitted to receive usual care including physical therapy and exercise and were not permitted to take analgesics and antiphlogistics during the periods.

INTERVENTIONS:
Device: Acupuncture — Tool : Acupuncture Seirin SJ 0.16 * 40 (mm) / SJ 0.18 * 50 (mm) L-type needles were used for the study.
  Made from stainless steel needle SEIRIN JAPAN
  Other Names: SEIRIN J-Type
  Arms: Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective and safe therapeutic method in the treatment of cervical pain, shoulder and upper extremity pain and discomfort due to Whiplash associated disorder. (Traumatic car accidents)

We recruit 40 participants who had cervical, shoulder and upper extremity pain and had discomfort due to Whiplash associated disorder. And then we check initial data of 40 participants (Pain;VAS, Cervical ROM, SF-36, SDS, CMI)

40 participants were randomly allocated to two groups ; acupuncture group or waiting-list group.

Acupuncture group: participants were given acupuncture treatment three times a week during 2 weeks, for 15 minutes at each session. After 6 times acupuncture treatments, we check information of participants again after 2 weeks(VAS, ROM, SF-36, SDS, CMI)

Waiting-list group : The waiting-list group did not receive acupuncture treatment. After 2 weeks we check information of participants again (VAS, ROM, SF-36, SDS, CMI)

The waiting-Patients in both groups were permitted to receive usual care including physical therapy and exercise and were not permitted to take analgesics and antiphlogistics during the trial periods.

DETAILED DESCRIPTION:
We recruited participants through advertisements in local newspapers or on the homepage of a Kyung-hee Medical Centre during December 8, 2009 to October 14, 2010.

Patients who met eligibility criteria were randomly allocated into either acupuncture treatment group or waiting-list group. Random sequences were generated by computerized number table. Allocation was concealed using sealed envelopes. According to priority, sealed envelope was matched when the patients had given informed consent.

The method of acupuncture: participants were given acupuncture treatment three times a week during 2 weeks, for 15 minutes (Needle retention time) at each session. (Total 6 times)

We select about ten acupuncture points

* Local Acupoints : SI14, SI15, BL10, BL12, BL13, BL14, TE15, GB20, SI9
* Distal Acupoints :

  * Upper extremities: LU6, LU7, LU9, LI11, HT3, SI2, SI3, SI5, SI7, PC4, PC6, TE5
  * Lower extremities: SP3, SP4, BL59, BL60, BL61, BL62, BL66, KI3, KI4,KI6, KI7, GB40, GB41, LR4

All Acupuncture points were prepared with 70% alcohol pads, and disposable stainless steel needles were used. Most of acupuncture were inserted vertically 1~2cm in depth until patient can feel De-Qi. (No more additional stimulation)

ELIGIBILITY:
Inclusion Criteria:

* The patients who suffer cervical pain, limitation of cervical ROM, discomfort sensation due to traffic accidents (Whiplash associated disorder)
* The patients who had no effect with 3 months orthopedical treatment.
* willing to give their permission approval.
* patients of at least 20 years of age (Both men, women)

Exclusion Criteria:

* Cervical fracture
* Cervical spondylosis
* suspect malignant disease(ex. tumor, stroke, etc)
* suspect hemorrhagic disease infection disease, inflammatory disease
* unable to communicate with Korean
* The patients who had conscious disorder
* Any other conditions deemed unsuitable for trial as evaluated by Physician-in-charge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | Change from Baseline in VAS at 2 weeks (post treatment)
  VAS which assessed the cervical and back pain intensity used a 0 to 10 point line, which zero corresponded to no pain and 10 to the extreme pain

SECONDARY OUTCOMES:
Cervical mobility on the Cervical ROM | Change from Baseline in cervical ROM at 2 weeks (post treatment)
  Cervical ROM was measured in six directions (Flexion, Extension, Right lateral bending, Left lateral bending, Right rotation, Left rotation) with goniometer.
Quality of life on the SF-36(36-Item Short-Form Health Survey) | Change from Baseline in SF-36 at 2 weeks (post treatment)
  SF-36, which assessed the quality of life, is composed of eight dimensions. Each dimension stands for Physical Functioning (PF), Social Functioning (SF), Role-Physical (RP), Bodily Pain (BP), Role-Emotional (RE), Mental Health (MH), Vitality (VT), General Health (GH)
SDS (Zung Self Rating Depression Scale) | Change from Baseline in SDS at 2 weeks (post treatment)
  SDS, the brief psychology examination consists of 20 questions, which each question has a 4-point rating scale (1 to 4) and sum score was multiplied 1.25 then total score varied from 25 to 100
CMI (Cornell Medical Index) | Change from Baseline in CMI at 2 weeks (post treatment)
  CMI, the brief psychology examination consists of eighteen section-195 questions. A to L section (144 questions) stands for physical state and M to R section (51 questions) stands for mental state. Answer 'yes' means that had a symptom and scores 2 point, and answer 'no' means that had not a symptom and score 1 point

CONTACTS AND LOCATIONS:
Overall Officials: Do Young Choi, Professor, Principal Investigator — Department of Acupuncture & Moxibustion, Kyunghee Oriental Medical Center.
Locations (1):
- Department of Acupuncture & Moxibustion, Kyunghee Oriental Medical Center, Seoul, Hoegi-dong, Dongdaemun-gu, Seoul, South Korea